CLINICAL TRIAL: NCT04698200
Title: Type 2 Diabetes, Cardiovascular Comorbidity and Environmental Temperature: Randomized Controlled Study
Brief Title: Type 2 Diabetes, Cardiovascular Comorbidity and Environmental Temperature
Acronym: DiabColdHeat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oulu (Other)
Collaborators: Finnish Institute of Occupational Health (Other); University of Texas Southwestern Medical Center (Other); Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DiabColdHeat
Record Dates: First submitted 2020-11-23; First posted 2021-01-06 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood pressure (Experimental): Measurement of brachial, central and beat-to-beat blood pressure.
  Interventions: Other: Cold exposure

INTERVENTIONS:
Other: Cold exposure — Whole body resting cold (+10 degrees centigrade) and heat (+40 degrees centigrade) for 60 minutes.
  Other Names: Heat exposure

SUMMARY:
Both high and low environmental temperatures are associated worldwide with higher morbidity and mortality and an estimated 8% of the mortality is estimated to relate to non-optimum temperatures. The majority of the adverse health effects occur at to low, and not high temperatures, and already with a modest change in temperature. Persons with type 2 diabetes can be sensitive to the effect of temperature due to their altered neural, metabolic and circulatory functions. The pathophysiological responses of type 2 diabetes in a cold and hot environment are not known.

The aim of the study is to examine how advanced type 2 diabetes (disease progression >10 years) alone, an in conjunction with coronary artery diseases and hypertension affect neural, cardiovascular and metabolic responses in a cold and hot environment.

Type 2 diabetes is associated with altered neural regulation, weakened cardiovascular function, structural changes in blood vessels, altered blood constitution and metabolic disturbances. These affect thermoregulation and result in increased susceptibility to cold (lesser heat production, increased heat loss) and heat (lesser sweating and heat loss).

The patients are exposed under controlled conditions in a random order to both cold (+10°C) and heat (+44°C) while resting and lightly clothed for 90 min at a time. The exposure itself is preceded by baseline measurements of the parameters of interest, and followed by repeating the same measurements after the exposure.

The topic of the research is very relevant due to the worldwide epidemic of type 2 diabetes. Simultaneously, the comorbid conditions associated with diabetes become more common and are related to a higher occurrence of cardiac events. The research information is useful for all individuals with type 2 diabetes in their protection and self-management of the disease, and enabling to maintain functional ability in a cold or hot environment. The research knowledge can be utilized when developing weather warning systems for the identification of susceptible populations. Health care personnel may utilize the research information while advising their patients and for proper care. An increased awareness of the health effects of both low and high temperatures improve the functional ability of individuals and reduced help reducing morbidity and mortality from weather conditions.

DETAILED DESCRIPTION:
Significance of the project in relation to current knowledge Temperature, health and climate change. Both high and low and environmental temperatures cause discomfort and degradation of physical performance. These normal physiological responses elicited to lose or preserve body heat can aggravate the course of chronic diseases and lead to a higher amount of health care visits, hospitalizations, or deaths. Globally, most of the adverse health effects are caused by cold, rather than heat, and occur already at mild non-optimal temperatures.

Environmental temperatures reflect the primary effects of climate change (CC), the biggest health threat of the 21st century. CC primarily involves a global increase of temperatures, and especially in the frequency, intensity and duration of heat extremes. Connected to the variability of weather, also higher amounts of precipitation, clouds, and winds are predicted. Northern climates, such as Finland, are subjects to huge annual variations in temperature (from ca. +30°C to -30°C) together with periodic prolongation of temperature extremes (heat and cold spells). Global projections predict that health effects of cold continue to outnumber those of heat in Finland, but heat exposure becomes increasingly important, also due to the lack of adaptation to high temperatures of northern residents.

T2D and temperature. The global occurrence of diabetes is 425 million people of which 77% are working aged and is estimated to increase to 629 million people by 2045. Type 2 diabetes (T2D) accounts for 90% of the diabetic patients. In Finland, the incidence of T2D has increased markedly in men for the last 35 years. Diabetes of all types can lead to micro- (retino-, nephro- and neuropathies) and macrovascular (cerebral, coronary and peripheral arterial disease) complications and resulting in higher morbidity and premature deaths. The economic burden of the direct and indirect costs of diabetes is tremendous and represented 1.8% of the GDP in 2015.

Epidemiological studies suggest that non-optimal environmental temperatures and diabetes are associated with higher morbidity and mortality. A study of 4.5 Million GP consultations showed that persons having T2D sought medical attention more often with both low and high temperatures. Furthermore, cold and hot temperatures were associated with a 12% and a 30% increase in diabetes-related hospitalizations.

Heat exposure may involve a lesser ability to lose additional body heat (higher heat load) to the environment and higher cardiovascular strain.

To our knowledge, there are only three controlled studies that have assessed whole-body heat exposure among persons with T2D. In healthy persons high temperatures dilates superficial blood vessels enabling conveying additional body heat to the environment. Consequently, blood flow is directed to the body surface augmenting heart rate and cardiac workload. In persons with T2D the dilation of the blood vessels may be delayed and lead to diminished capacity to lose heat through skin circulation. In addition, disrupted endothelial function and stiffening of blood vessels can lead to an attenuated reduction in blood pressure. Factors, such as reduced sweating capacity, as well as autonomic and peripheral neuropathies may further impair the ability to lose body heat to the environment. In fact, a study involving older adults with T2D detected reduced capacity to lose additional body heat during exercise, resulting in greater thermal strain. Also, cardiac regulation and ability to increase cardiac workload could be impaired in T2D under exposure to heat. Supporting this, older (ca. 60 yrs.) persons with T2D showed reduced heart rate variability and response to heat. Lastly, hypercoagulation of persons with T2D could be further increased during heat exposure, but there are no studies of the topic.

Cold exposure may involve higher cardiovascular strain and a reduced ability to produce or preserve (increased heat loss) body heat in cold weather in persons with T2D.

There are no previous controlled studies which assess the effects of whole-body cold exposure among persons with T2D. In healthy persons exposure to low temperature increases sympathetic activity which constricts superficial blood vessels, results in elevated blood pressure and cardiac workload. The aggravated blood pressure increase in persons with T2D can be due to sympathetic over activity, disrupted endothelial function and stiffer arteries. The altered neural regulation in T2D may impair cardiac responsiveness to the higher cardiac workload and oxygen demand in cold. Cold exposure also increase blood coagulation potential, which together with hypercoagulability related with T2D, could promote the production of thromboses and adverse cardiac events. Microvascular dysfunction associated with autonomic neuropathy can also impair vascular responsiveness during local cooling and possibly increase susceptibility to low temperatures. Cold exposure may also be related to reduced heat production (shivering thermogenesis or reduction in brown adipose tissue activity and mass).

Modifying factors possibly affecting vulnerability to high or low temperature of T2D High blood pressure is reported in over two-thirds of patients with T2D and the incidence of diabetes and hypertension (HTN) predicts each other over time. The two diseases share common metabolic abnormalities and insulin resistance is a characteristic of both prediabetes and prehypertension. Like diabetes, also cardiovascular diseases are temperature sensitive. Glycemic control may be important for coping with thermal stress, but the available evidence is scarce. Heat exposure, especially when combined with exercise, can induce hypoglycemia. On the other hand, a brief acclimation period to repeated mild cold exposure can improve insulin sensitivity and glycemic state. Medication associated with both treatment of T2D itself (metformin, gliptines, gliflotsines) or HTN (beta-blockers, diuretics, calcium-channel blockers, ACE-inhibitors), could significantly affect cardiovascular and thermal responses, but their association with health outcomes are not known. Regular physical activity itself reduces HbA1c, but may also improve heat dissipation capacity, but the mechanisms are unclear.

Our aims are:1) Assess how advanced T2D in combination with hypertension, influences cardiovascular function and associated neural, and metabolic responses during whole-body passive exposure to heat (activating heat loss through higher superficial circulation and sweating) and cold (causing increase in heat production and reduction in superficial circulation) and compared with healthy persons. 2) Eamine how different diabetic micro- and macrovascular complications involving varying degrees of severity, affect the observed cardiovascular, neural and metabolic functions while exposed to either cold or heat. 3) Assess how T2D (diagnosed or detected during clinical examination) alone, and in combination with hypertension (diagnosed or measured during clinical examination) affect reported cold- or heat-related cardiorespiratory symptoms and consequently, from a longitudinal perspective, hospitalizations and mortality. We also aim to identify the influence of potential determinants, such as the use of medication, physical activity and other demographic, socioeconomic and lifestyle factors.

Research hypotheses: 1) Exposure of those with T2D may lead to earlier heat strain due to reduced ability to lose (reduced sweating and circulation) bodily heat at high temperatures. 2) Exposure to cold may lead to earlier cold strain due to weakened ability to preserve (impaired circulation) or produce bodily heat (shivering) at low temperatures. 3) Having more complications increase the vulnerability to these environments. 4) At the population level, people with T2D report more heat- and cold-related cardiorespiratory symptoms and experience more hospitalizations and deaths. These effects are dependent on the glycemic and blood pressure control, use of medication and other lifestyle factors. 5) Health care visits and mortality are preceded by temperatures that are higher or lower than average.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Type 2 diabetes
* Hypertension

Exclusion Criteria:

* Smoking
* Chronic respiratory diseases
* Coronary artery diseases

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change of systolic and diastolic blood pressure | 10, 20 and 30 minutes before the intervention, during the intervention in 10 minutes intervals, and 5, 10, 15, 20 25 and 30 minutes after the intervention.
  Brachial, central and beat-to-beat systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Electrocardiogram, ECG | 3 hours
  Continuous 15-channel recording during the intervention to detect ST elevation.
Metabolic rate | During the 60 minutes intervention period.
  Measurement of oxygen consumption.
Sweating | During the 60 minutes intervention period and immediately after the intervention.
  Measurement of total sweating rate.
Skin and body temperature | 3 hours
  Continuous measurement of skin and body temperatures.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oulu, Center for Environmental and Respiratory Health Research, Oulu, Finland